CLINICAL TRIAL: NCT01929486
Title: Phase Ia/Ib Multicenter Trial of Mogamulizumab for Advanced or Recurrent Cancer.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aichi Medical University (Other)
Responsible Party: Principal Investigator, Ryuzo Ueda, MD, Aichi Medical University, Aichi Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KW0761-IIT-01
Record Dates: First submitted 2013-07-24; First posted 2013-08-28 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Solid Tumor
MeSH Terms: interventions — mogamulizumab

ARMS (3):
- <Phase Ia> Mogamulizumab 0.1mg/kg, 0.5mg/kg or 1.0mg/kg (Experimental): <Phase Ia> Dose-escalation method with Mogamulizumab 0.1mg/kg, 0.5mg/kg or 1.0mg/kg. Mogamulizumab will be administered 8 times every week.
  Interventions: Biological: Mogamulizumab
- <Phase Ib> Mogamulizumab of the tolerated dose (Experimental): <Phase Ib> Mogamulizumab of the tolerated dose in Phase Ia will be administered 8 times every week.
  Interventions: Biological: Mogamulizumab
- <Phase Ib> Mogamulizumab 0.1mg/kg (Experimental): <Phase Ib> Mogamulizumab 0.1mg/kg will be administered 8 times every week.
  Interventions: Biological: Mogamulizumab

INTERVENTIONS:
Biological: Mogamulizumab — Mogamulizumab 0.1mg/kg, 0.5mg/kg or 1.0mg/kg will be administered 8 times every week.
  Other Names: KW-0761

SUMMARY:
The purpose of this study is to investigate safety, pharmacokinetics, effect of regulatory T cell depletion with Mogamulizumab for advanced or recurrent cancer patients.

DETAILED DESCRIPTION:
This study consists of phase Ia and Ib portions for patients with solid tumors.

Phase Ia portion is the standard 3+3 dose-escalation design with 0.1mg/kg, 0.5mg/kg and 1.0mg/kg of Mogamulizumab.

Phase Ib portion is the randomized study comparing 0.1mg/kg and tolerated dose of Mogamulizumab based on the phase Ia portion to pursue safer and immunologically more efficient dose.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed, CCR4 negative lung, stomach, esophageal, ovarian or skin cancer.
2. Patients with therapy-resistant cancer. Patients with recurrent cancer or advanced cancer who refused standard therapies.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status is 0, 1 or 2.
4. Patients should be 20 years or older at the time of informed consent.
5. No serious dysfunction of major organs (bone marrow, heart, lung, liver and kidney) and meet the following conditions ; 1) WBC count : >=1,500/mm3 2) Hemoglobin : >=8.0g/dL 3) Platelet count : >=75,000/mm3 4) Serum total bilirubin : <=2.0 x ULN 5) AST and ALT : <=2.5 x ULN (Patients with hepatic infiltration which is attributed to primary disease<=5.0 x ULN) 6) Serum creatinine : <=1.5 mg/dL 7) SpO2 : >=93 % 8) ECG : No abnormal findings. 9) EF : >=50 %
6. Agree to use birth control including condom etc. from the time of obtaining the first consent to 24 weeks after the final administration of the study drug (except female after menopause (1 year or more after the last menstruation) and female/male after the operation for sterilization).
7. Given written informed consent.
8. Patients who can be hospitalized from the day of first administration to the next day.
9. Patients who have target lesions measurable by RECIST ver.1.1.
10. Life expectancy >= 3 months.

Exclusion Criteria:

1. Patients with HIV antibody positive.
2. Patients with HCV antibody positive.
3. Patients with autoimmune disease.
4. Patients with HBs antigen or HBV-DNA positive.
5. History of serious anaphylaxis induced by antibody preparation.
6. Patients with double cancer.
7. Within 4 weeks after treatment with anticancer agent, immune suppressant, immune enhancer, cytokine therapy, radiotherapy or surgery for the primary disease.
8. Pregnant or breast-feeding females and females who have a possibility of pregnancy.
9. Patients with active infection.
10. Patients with psychosis or dementia.
11. Patients who need continuous systemic administration of adrenocorticosteroid.
12. Patients who have received hematopoietic stem cell transplantation.
13. Patients who have presence or suspicion of CNS involvement.
14. Patients who are administered the other investigational product within 4 weeks of the entry.
15. Patients treated with immunotherapy for cancer (e.g. cancer vaccine therapy) within 12 weeks of the entry.
16. Any other inadequacy for this study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2013-02; Primary Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose(MTD) of Mogamulizumab | from first administration until day 28
Dose limiting toxicity(DLT) of Mogamulizumab | from first administration until day 28
Number of adverse events | from first administration to 24 weeks after the final administration, an expected average of 32 weeks.
Cmax of Mogamulizumab | from day 0 to 28 days after the final administration, an expected average of 12 weeks.
Ctrough of Mogamulizumab | from day 0 to 28 days after the final administration, an expected average of 12 weeks.
AUC0-7day of Mogamulizumab | from day 0 to 28 days after the final administration, an expected average of 12 weeks.
Rate of Treg decrease in PBMC compared to baseline | from baseline to every 4 weeks until data cut off

SECONDARY OUTCOMES:
Objective tumor response rate according to RECIST | from baseline to every 12 weeks, until data cut off
Median progression free survival rate | from baseline to every 12 weeks, until data cut off (expected date is March 2016)
Median Overall survival rate | from baseline to every 12 weeks, until data cut off

CONTACTS AND LOCATIONS:
Locations (1):
- Aichi Medical University, Nagoya, Aichi-ken, Japan

REFERENCES:
- [Derived] Fujikawa K, Saito T, Kurose K, Kojima T, Funakoshi T, Sato E, Kakimi K, Iida S, Doki Y, Oka M, Ueda R, Wada H. Integrated analysis of phase 1a and 1b randomized controlled trials; Treg-targeted cancer immunotherapy with the humanized anti-CCR4 antibody, KW-0761, for advanced solid tumors. PLoS One. 2023 Sep 20;18(9):e0291772. doi: 10.1371/journal.pone.0291772. eCollection 2023. PMID 37729184
- [Derived] Maeda Y, Wada H, Sugiyama D, Saito T, Irie T, Itahashi K, Minoura K, Suzuki S, Kojima T, Kakimi K, Nakajima J, Funakoshi T, Iida S, Oka M, Shimamura T, Doi T, Doki Y, Nakayama E, Ueda R, Nishikawa H. Depletion of central memory CD8+ T cells might impede the antitumor therapeutic effect of Mogamulizumab. Nat Commun. 2021 Dec 14;12(1):7280. doi: 10.1038/s41467-021-27574-0. PMID 34907192